CLINICAL TRIAL: NCT05024240
Title: Interaction of the Cognitive and Sensory-cognitive Tasks With Postural Stability in Individuals With Stability Disorders Based on Cerebellar Ataxia
Brief Title: Interaction of the Cognitive and Sensory-cognitive Tasks With Postural Stability in Individuals With Stability Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Mgr. Kateřina Levínská, principal investigator, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: ID 14827
Record Dates: First submitted 2021-08-11; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Cerebellar Ataxia; Cerebellar Diseases
Keywords: Stability; Dual Task; Cerebellum; Stroop Test; Backward Counting Test
MeSH Terms: conditions — Cerebellar Ataxia; Cerebellar Diseases

STUDY DESIGN:
Intervention Model Description: There will be group of patients with disorders od cerebellum and control group of healthy age-matching probands
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient group (Experimental): 20 patients with cerebellum disorders, who suffer from stability disorders and with specific 3 Hz tremor
  Interventions: Diagnostic Test: Stabilometry; Diagnostic Test: Stroop test; Diagnostic Test: Backward counting test
- Control group (Active Comparator): 20 healthy age-matching probands without any neurological disorders and stability issues
  Interventions: Diagnostic Test: Stabilometry; Diagnostic Test: Stroop test; Diagnostic Test: Backward counting test

INTERVENTIONS:
Diagnostic Test: Stabilometry — Probands will stand on stabilometric platform (double leg stance) and we will measure CoP parameters area and length. We also make this task harder by using foam and exclusion of visual control. Length of one test is 30s.
Diagnostic Test: Stroop test — There are various names of colours written in non-matching font colour in this test. During this test probands are required to name the colour which is written in text not the colour of the font. We will measure reaction time and number of mistakes.
Diagnostic Test: Backward counting test — In this counting test probands are given number from interval <180-200> and they are asked to subtract 7 during 30s interval of the testing. We will measure reaction time and number of mistakes.
  Other Names: BCT

SUMMARY:
The aim of this study is to describe the interaction of the cognitive and visual-cognitive task with postural stability in patients suffering by cerebellar ataxia. Investigators will measure changes in postural stability parameters and in secondary task performance, which should show the ability of the patients to manage the dualtask situations.

DETAILED DESCRIPTION:
The aim of this research will be to describe the interaction between cognitive and cognitive sensory tasks and stability in patients whose disease impairs the ability to maintain a stable upright position, for example in patients with cerebellar syndromes. And further compare this interaction with a control group of healthy probands. This interaction will be investigated in variously demanding postural situations (eg. standing on both lower limbs, with the exclusion of visual control, with reduced proprioceptive input from the patch).

Patient stability will be quantified using a stabilometric examination on the Kistler platform (Kistler Instrumente AG, Switzerland). investigators will quantify the performance of patients in secondary tasks using parameters such as response time to response and success in assigned tests.

The expected number of probands is 20 individuals in both groups. Study will objectify postural stability by means of a static stabilometric examination on the Kistler platform, the recording length of each postural situation will be 30 s. Four different demands of postural tasks were chosen - a bipedal stand, a bipedal stand with the exclusion of visual control, a stand on a foam pad and a stand on a foam pad with the exclusion of visual control. To evaluate postural deviations, investigators chose the following CoP parameters: stabilogram curve length and stabilogram area. During the stabilometric measurement, the number of touches of the guardrail will also be recorded, or the number of falls or touches with a lightened limb of the pad or the other limb during the measurement. Testing will take place in the Neurological Laboratory of the Department of Neurology, 2nd Faculty of Medicine, Charles University in Prague and FN Motol.

Gradually, two types of secondary task will be added to the postural tasks, with visual input (modified Stroop test) and a purely cognitive task (Backward counting test). At first, probands will be acquainted with what types of tasks await them during the experiment and will be able to train each of them in two trial experiments. This will be followed by testing trials in random order (cognitive tests in single-task situations, namely sitting in a chair, single task postural tasks and dual-task situations).

ELIGIBILITY:
Inclusion Criteria:

* 3 Hz tremor in in frequency analysis (posturografy)
* stability disorder caused by cerebellar disorders in diagnose

Exclusion Criteria:

* lower than high school education
* vestibular disorders
* ankle instability
* other specific stability disorders
* unability to stand for 30s

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Centre of pressure - AREA (mm2) | 1 week
  the area below the graph of the curve formed by the movement of the patient's center of gravity during the 30 seconds while standing on the platform, computer processed (Kistler programme), measured in squared millimeters
Centre of pressure - LENGHT (mm) | 1 week
  the length of the curve formed by the movement of the patient's center of gravity during 30 seconds while standing on the platform, computer processed (Kistler programme), measured in millimeters
Reaction time in secondary tasks (ms) | 1 week
  time (measured in milliseconds) between individual responses of probands in a cognitive or visual test, measured from an audio recording of proband´s responses using a professional audio editing program

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Kolář, Prof. PaedDr. Ph.D., Study Chair — Department of Rehabilitation and Sports Medicine, Second Faculty of Medicine, Charles University; Ondřej Čakrt, Doc. PhDr. Ph.D., Study Director — Department of Rehabilitation and Sports Medicine, Second Faculty of Medicine, Charles University; Kateřina Levínská, Mgr., Principal Investigator — Department of Rehabilitation and Sports Medicine, Second Faculty of Medicine, Charles University
Locations (1):
- Second Faculty of Medicine, Charles University, Prague, Czechia